CLINICAL TRIAL: NCT00188864
Title: Dexamethasone as Palliative Treatment in Addition to Radiation Therapy for Patients With Brain Metastases: A Prospective Study
Brief Title: Dexamethasone for Palliation - Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 03-0662-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Dexamethasone

INTERVENTIONS:
Drug: dexamethasone

SUMMARY:
Brain metastases occur when cancer cells from the initial tumour site (for example, lung or breast) spread to the brain. This develops in approximately 10% - 30% of adults with cancer. They can produce different complaints related to their effect on brain functioning, decrease in a person's ability to carry on with their usual activities, a reduction in the quality of life and shortened life expectancy.

The standard treatment particularly for people with more than one brain metastasis consists of palliative radiation therapy to the brain and steroids. Steroids (such as Decadron or Dexamethasone) are medication used to reduce swelling around the tumour, and thus symptoms improve. Steroids could be very helpful but have a number of potential side effects, particularly if used for longer periods of time. There is no standard dose of Decadron used in treating brain metastases patients. The most commonly dose used is 4 mg four times/day.

This study will assess if lower doses of Decadron - 8 mg every morning for symptomatic patients and 4 mg every morning for asymptomatic patients - are effective in maintaining symptom control in patients with brain metastases, without neurological deterioration that necessitates the patient to go back or to a higher dose at any time. This information will help also in understanding how to decrease the side effects associated with higher doses of steroids in people with your condition.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of cancer (even if primary unknown)
* Brain metastases (single or multiple) confirmed by imaging (CT, MRI)
* No contraindication for RT/steroids
* Patient will be treated with Whole Brain Radiation Therapy
* Informed consent

Exclusion Criteria:

* Primary cancer is lymphoma or leukemia
* Complete surgical excision of brain metastases
* Patient was on steroids for more then 2 weeks prior to entering the study
* Confusion or other factors that would impair ability to assess symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-11; Primary Completion 2006-11 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
To perform an adequate statistical evaluation of patients regarding the role of steroid therapy in managing patients with cerebral metastases.

SECONDARY OUTCOMES:
To observe whether DXM 8mg qAM for symptomatic patients and DXM 4mg qAM for asymptomatic patients is effective in maintaining symptom control without neurological deterioration that necessitates the patient to go back to a higher dose.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bezjak, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada